CLINICAL TRIAL: NCT03152136
Title: A Pilot Study to Evaluate the Safety and Initial Effectiveness of the Cala ONE Device to Repeatably Aid in the Symptomatic Relief of Essential Tremor
Brief Title: A Pilot Study of the Cala ONE Device for Essential Tremor
Acronym: EXCITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cala Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ET-13
Record Dates: First submitted 2017-05-07; First posted 2017-05-12 (Actual); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: The first two weeks are a 3-arm parallel design (treatment, sham, and 'no intervention'). The second two weeks are open-label (all subjects cross-over to treatment arm).
Who Masked: Participant, Outcomes Assessor
Masking Description: The first two weeks of the study are double-blinded for the treatment and sham arms. The subjects and rating movement disorder neurologists will be blinded to the therapy allocation for the treatment and sham arms. The subjects in the 'no intervention' arm and their rating neurologists will not be blinded to their therapy allocation.
  The last two weeks are open-label, and all subjects will be given the option to use the Cala ONE device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- TAPS (Experimental): Subjects will receive a Cala ONE device that delivers TAPS, transcutaneous afferent patterned stimulation.
  Interventions: Device: Cala ONE device
- Sham (Sham Comparator): Subjects will receive a Cala ONE device that delivers sham stimulation.
  Interventions: Device: Cala ONE device
- No Intervention (No Intervention): Subjects will not receive a Cala ONE device, and will stay on their current treatment regimen for their essential tremor.

INTERVENTIONS:
Device: Cala ONE device — The Cala ONE device is a wrist-worn stimulator which applies a tremor-customized stimulation pattern to an individual's nerves.
  Arms: Sham; TAPS

SUMMARY:
Prospective, multi-center, randomized, controlled study designed to evaluate safety and repeatable effectiveness. Subjects will be randomized 2:1:1 to transcutaneous afferent patterned stimulation (TAPS), sham, or 'no intervention', respectively. Subjects randomized to the TAPS and sham arms will be blinded to their randomization assignments for the first two weeks of participation (controlled phase). After the first two weeks, all subjects will be crossed over to TAPS (open-label phase) for 2 weeks. During study participation, all subjects are to remain on a stable dosage of medications prescribed for the treatment of essential tremor, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥22 and ≤80 years of age
* Competent and willing to provide written, informed consent to participate in the study
* A diagnosis of essential tremor as confirmed from clinical history and examination by a movement disorder neurologist
* Postural, action or intention tremor severity score of 2 or above in the dominant hand/arm as measured by the CRST rating scale
* Significant disability due to essential tremor (Bain & Findley score of 3 or above in any one of the hand items)
* Currently or previously prescribed either propranolol or primidone for the treatment of essential tremor
* Stable dose of tremor medications for 30 days prior to study entry
* Stable dose of antidepressant medications for 90 days prior to study entry
* Willing to comply with study protocol requirements including: remaining on a stable dosage of tremor and antidepressant medications, if applicable, during the duration of the study; no significant alcohol or caffeine consumption within 12 hours of study visits; and no significant alcohol or caffeine consumption within 4 hours of twice-daily at home assessments during the controlled phase of the study

Exclusion Criteria:

* Moderate to severe ethanol dependence as defined by the criteria outlined in the DSM-5 (score of 4 or higher)
* Implanted electrical medical device, such as a pacemaker, defibrillator, or deep brain stimulator
* Previous thalamotomy procedure, including stereotactic thalamotomy, gamma knife radiosurgical thalamotomy, and focused ultrasound for the treatment of tremor
* Suspected or diagnosed epilepsy or other seizure disorder
* Swollen, infected, inflamed areas, or skin eruptions, open wounds, or cancerous lesions of skin at stimulation site
* Peripheral neuropathy affecting the tested upper extremity
* Presence of any other neurodegenerative disease like Parkinson-plus syndromes suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and Alzheimer's disease.
* Anyone suspected to have the diagnosis of idiopathic Parkinson's disease (PD). This includes excluding anyone with the presence of parkinsonian features including bradykinesia rigidity, or postural instability. Subjects who exhibit only mild resting tremor but no other symptoms or signs of PD may be included.
* Botulinum toxin injection for hand tremor within 6 months prior to study enrollment
* Are participating or have participated in another interventional clinical trial in the last 30 days which may confound the results of this study, unless approved by the Sponsor
* Are participating or have participated in another Cala Health clinical trial
* Significant alcohol or caffeine consumption within 12 hours of study enrollment, which may confound the results of the study, where significant caffeine is considered more than 95 mg (equivalent to a cup of coffee), and significant alcohol is considered more than 14 g (equivalent to 5 oz of wine, 12 oz of beer, or 1.5 oz of distilled spirits).
* Subjects unable to communicate with the investigator and staff
* Any health condition that in the investigator's opinion should preclude participation in this study
* Pregnancy or anticipated pregnancy during the course of the study

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Personal Care Neurology, Oakland, California
  - Movement & Neuroperformance Center, Denver, Colorado
  - Kansas University Medical Center, Kansas City, Kansas
  - EvergreenHealth, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No
Data will be published, but no PHI will be made available.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAPS | Sham | No Intervention
Started | 32 | 15 | 15
Completed | 29 | 15 | 14
Not Completed | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAPS | Sham | No Intervention | Total
Number analyzed (Participants) | 32 | 15 | 15 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (8) | 66 (11) | 67 (9) | 67 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 7 | 6 | 34
  Male | 11 | 8 | 9 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 31 | 15 | 15 | 61
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 30 | 15 | 15 | 60
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 15 | 15 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Tremor Power
Description: For TAPS and sham arms, subjects will be prompted to perform a lateral postural hold prior to entering their PGI-S score before and after each stimulation session. During this hold, the device will record motion data to objectively assess if there are any changes in tremor level.
Time Frame: Mean tremor power pre stimulation over two weeks of device usage as compared to mean tremor power post stimulation over two weeks of device usage.
Measure: Mean (Standard Deviation); unit: percent tremor improvement
Arm/Group | TAPS | Sham
Number analyzed (Participants) | 29 | 14
percent tremor improvement | 43 (4) | 9 (10)

2. Other Pre Specified Outcome: Change in Clinical Rating Scale for Tremor (CRST) After Stimulation
Description: A complete CRST examination (also known as the Fahn-Tolosa-Marin Tremor Rating Scale) will be completed at baseline for all arms: TAPS, sham, and 'no intervention.' For TAPS and sham arms, a subset of CRST relevant to upper limb tremor will be repeated after stimulation.
Time Frame: Collected before and after in-office stimulation sessions at Week 2
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Change in Clinical Global Impression of Severity (CGI-S)
Description: Tremor severity will be assessed with the 7-point CGI-S scale at baseline for all arms. For TAPS and sham arms, CGI-S will also be assessed during and after stimulation.
Time Frame: Collected before, during, and after in-office stimulation sessions at Week 0, Week 2, and Week 4
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Clinical Global Impression of Improvement (CGI-I)
Description: For TAPS and sham arms, the blinded rating neurologist will assess improvements in tremor level during and after stimulation.
Time Frame: Collected during and after in-office stimulation sessions at Week 0, Week 2, and Week 4
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Bain & Findley Activities of Daily Living (ADL) Scale
Description: The complete Bain & Findley ADL questionnaire will be administered at baseline for all arms. For TAPS and sham arms, a subset of ADLs relevant to upper limb tremor will be repeated with provided props during and after stimulation.
  On a weekly basis, all subjects will answer the complete Bain & Findley ADL questionnaire via phone call.
Time Frame: Collected before, during, and after in-office stimulation sessions at Week 0, Week 2, and Week 4. Collected via phone call Week 1 and Week 3.
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Subject Impression of Durability of Effect
Description: TAPS and sham arms will also be asked how long their tremor relief lasts due to stimulation, if applicable.
Time Frame: Week 1, 2, 3 and 4.
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Quality of Life in Essential Tremor Questionnaire (QUEST)
Description: The QUEST assessment will be administered to all subjects during in-office visits (every 2 weeks).
Time Frame: Week 0, 2, and 4
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Patient Global Impression of Severity (PGI-S)
Description: Tremor severity will be assessed with the 7-point PGI-S scale at baseline for all arms. For TAPS and sham arms, PGI-S will also be assessed during and after stimulation during office visits.
  Additionally, for TAPS and sham arms, PGI-S will be entered on the device before and after each stimulation session in the home environment.
Time Frame: Before and after every stimulation session for TAPS and sham subjects through study completion. Twice daily for 'no intervention' subjects through study completion.
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Patient Global Impression of Improvement (PGI-I)
Description: For TAPS and sham arms, the blinded subject will assess improvements in their tremor level during and after stimulation during office visits.
Time Frame: Collected during and after in-office stimulation sessions at Week 0, Week 2, and Week 4
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Subject Survey of Satisfaction
Description: At the final visit, all subject will take a subject satisfaction survey which will include questions such as likelihood to recommend and other questions related to the usability of the device.
Time Frame: Week 4
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Device Usage Metrics
Description: For TAPS and sham arms, the device will record usage metrics such as how many times the device was used per day and stimulation amplitude, to assess if there are any changes over time within group and within subject.
Time Frame: Week 4
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Clinical Rating Scale for Tremor (CRST) After Stimulation
Description: as for outcome 2
Time Frame: Collected before and after in-office stimulation sessions at Week 0 and 4.
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Clinical Rating Scale for Tremor (CRST) During Stimulation
Description: A complete CRST examination (also known as the Fahn-Tolosa-Marin Tremor Rating Scale) will be completed at baseline for all arms: TAPS, sham, and 'no intervention.' For TAPS and sham arms, a subset of CRST relevant to upper limb tremor will be repeated during stimulation.
Time Frame: Collected before and during in-office stimulation sessions at Week 0, 2 and 4.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | TAPS | Sham | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 5/32 | 1/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAPS (N=32) | Sham (N=15) | No Intervention (N=15)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Discomfort (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT03152136/Prot_000.pdf